CLINICAL TRIAL: NCT06374576
Title: Improving EHealth Literacy of Older Adults in Hong Kong: a Randomized Controlled Trial Study
Brief Title: Improving EHealth Literacy of Older Adults in Hong Kong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Sino Group (Unknown); NG TENG FONG Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCIEL
Record Dates: First submitted 2024-04-09; First posted 2024-04-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: EHealth Literacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lecture on eHealth literacy and digital intervention (Experimental): Participants in the intervention group will receive a health promotion education program for improving eHealth literacy. The education program will include a 1.5-hour lecture and a 1-week digital intervention
  Interventions: Behavioral: Lecture on eHealth literacy; Behavioral: Digital intervention on eHealth literacy
- Lecture on general health and digital intervention (Placebo Comparator): Participants in the control group will receive a health promotion education program about general health. The education program will include a lecture and a 1-week digital intervention
  Interventions: Behavioral: Lecture on general health; Behavioral: Digital intervention on general health

INTERVENTIONS:
Behavioral: Lecture on eHealth literacy — There will be a lecture on eHealth literacy. The lecture will be delivered by one well-trained lecturer. , the lecture will be held for old adults in small groups, including a structured curriculum consisting of 4 parts: 5 minutes for the introduction, 40 minutes for the lecture and demonstration, and 40 minutes for hands-on session, 5 minutes for wrapping up. The contents covered in the 40-minute lecture were as follows: 1) smartphone internet basics; 2) introduction of the website prepared for this study; 3) evaluation of the credibility of online health information.
  Arms: Lecture on eHealth literacy and digital intervention
Behavioral: Digital intervention on eHealth literacy — 1-week digital intervention, which are multiple messages about the lecture topic will be provided
  Arms: Lecture on eHealth literacy and digital intervention
Behavioral: Lecture on general health — A lecture session that focus on the general health but not eHealth literacy will be provided
  Arms: Lecture on general health and digital intervention
Behavioral: Digital intervention on general health — 1-week digital intervention, which are multiple messages about the lecture topic will be provided
  Arms: Lecture on general health and digital intervention

SUMMARY:
This study is an randomized controlled trial (RCT) study to examine the feasibility and effectiveness of a community-based health promotion education intervention for improving the eHealth literacy of older adults

DETAILED DESCRIPTION:
Background: Potential positive health outcomes were related to improved eHealth literacy. It is crucial to identify the population groups that may have low eHealth literacy. This eHealth literacy trail aims to design health promotion education intervention to improve the eHealth literacy of older adults in Hong Kong.

Study design: This RCT study will be conducted at the local non-governmental organization (NGO) centers in Hong Kong. Participants in the intervention group will receive a health promotion education program for improving eHealth literacy. The education program will be delivered through collaborative learning, including a 1.5-hour lecture and a 1-week digital intervention

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years old or above
* Smartphone user
* Reported lower eHealth literacy scores (eHEALS < 26) in previous study

Exclusion Criteria:

* All subjects have the right to withdraw if they wish not to continue

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
eHealth literacy | Baseline, 2-week, 3- and 6-month after intervention
  eHealth literacy score will be assessed with the 8-item eHealth literacy Scale (eHEALS) on a five-point Likert scale. The scale range from 8 to 40, higher scores means a better e-health literacy.

SECONDARY OUTCOMES:
Health Knowledge Learning Intention | Baseline, 2-week, 3- and 6-month after intervention
  To measure the health knowledge learning intention, the three-item questionnaire were adopted and modified from existing studies. This is a five-point Likert scale ranging from 3 to 15, with higher scores means higher health knowledge learning intention.
Online Health Information Seeking | Baseline, 2-week, 3- and 6-month after intervention
  Modified from the measurement adopted and revised from existing study, three-item questionnaire were used to test online health information-seeking behavior. This is a five-point Likert scale ranging from 3 to 15, with higher scores means better online health information seeking.
Online Health Information Scanning | Baseline, 2-week, 3- and 6-month after intervention
  Three-item questionnaire borrowed from existing studies were developed to measure online health information-scanning behavior. This is a five-point Likert scale ranging from 3 to 15, with higher scores means better online health information scanning.
Health-promotion behaviors | Baseline, 2-week, 3- and 6-month after intervention
  To measure health-promotion behaviors, 24 questions were developed adopted from existing studies, which contains six dimensions (Exercise, Nutrition, Self-actualization, Interpersonal Support, Health Responsibility, Stress Management), with a 4-item sub-scale allocated to each dimension. For each sub-scale, this is a four-item Likert scale ranging from 4 to 16, with higher scores means better outcome in this dimension.
Health Decision Change | Baseline, 2-week, 3- and 6-month after intervention
  Health Decision Change. Measurements of health decision change were adapted and modified from existing studies. A total of three items are developed to measure older adults' health decision change based on the health information acquired from their smartphones. This is a five-point Likert scale ranging from 3 to 15, with higher scores means greater health decision change .

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berkowsky RW. Exploring Predictors of eHealth Literacy Among Older Adults: Findings From the 2020 CALSPEAKS Survey. Gerontol Geriatr Med. 2021 Dec 14;7:23337214211064227. doi: 10.1177/23337214211064227. eCollection 2021 Jan-Dec. PMID 34926723
- [Background] Pourrazavi S, Kouzekanani K, Bazargan-Hejazi S, Shaghaghi A, Hashemiparast M, Fathifar Z, Allahverdipour H. Theory-based E-health literacy interventions in older adults: a systematic review. Arch Public Health. 2020 Aug 10;78:72. doi: 10.1186/s13690-020-00455-6. eCollection 2020. PMID 32793345
- [Background] Xie B. Effects of an eHealth literacy intervention for older adults. J Med Internet Res. 2011 Nov 3;13(4):e90. doi: 10.2196/jmir.1880. PMID 22052161
- [Background] Chang SJ, Yang E, Lee KE, Ryu H. Internet health information education for older adults: A pilot study. Geriatr Nurs. 2021 Mar-Apr;42(2):533-539. doi: 10.1016/j.gerinurse.2020.10.002. Epub 2020 Oct 19. PMID 33092906
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046
- [Background] Wong DK, Cheung MK. Online Health Information Seeking and eHealth Literacy Among Patients Attending a Primary Care Clinic in Hong Kong: A Cross-Sectional Survey. J Med Internet Res. 2019 Mar 27;21(3):e10831. doi: 10.2196/10831. PMID 30916666
- [Background] Waters EA, Wheeler C, Hamilton JG. How Are Information Seeking, Scanning, and Processing Related to Beliefs About the Roles of Genetics and Behavior in Cancer Causation? J Health Commun. 2016;21(sup2):6-15. doi: 10.1080/10810730.2016.1193917. Epub 2016 Sep 23. PMID 27661291
- [Background] Zhang L, Jung EH, Chen Z. Modeling the Pathway Linking Health Information Seeking to Psychological Well-Being on WeChat. Health Commun. 2020 Aug;35(9):1101-1112. doi: 10.1080/10410236.2019.1613479. Epub 2019 May 15. PMID 31088169
- [Background] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262
- [Background] Ruggiero KJ, Gros DF, McCauley J, de Arellano MA, Danielson CK. Rural adults' use of health-related information online: data from a 2006 National Online Health Survey. Telemed J E Health. 2011 Jun;17(5):329-34. doi: 10.1089/tmj.2010.0195. Epub 2011 Apr 27. PMID 21524201
- [Background] Fisher WA, Fisher JD, Harman J. The information-motivation-behavioral skills model: A general social psychological approach to understanding and promoting health behavior. In: Social Psychological Foundations of Health and Illness. Malden, MA, USA: Blackwell Publishing Ltd; 2010. p. 82-106.
- [Background] Shang L, Zuo M. Investigating older adults' intention to learn health knowledge on social media. Educ Gerontol [Internet]. 2020;46(6):350-63.
- [Background] Ahadzadeh AS, Pahlevan Sharif S, Sim Ong F. Online health information seeking among women: the moderating role of health consciousness. Online Inf Rev [Internet]. 2018;42(1):58-72.
- [Background] Wei MH, Lu CM. Development of the short-form Chinese health-promoting lifestyle profile. J Health Educ. 2005;24:25-46.
- [Background] Song J, Li Y, Guo X, Shen KN, Ju X. Making mobile health information advice persuasive: An Elaboration Likelihood Model perspective. J Organ End User Comput [Internet]. 2022;34(4):1-22.